CLINICAL TRIAL: NCT04380935
Title: Effectiveness and Safety of Convalescent Plasma Therapy on COVID-19 Patients With Acute Respiratory Distress Syndrome in Referral Hospitals in Indonesia
Brief Title: Effectiveness and Safety of Convalescent Plasma Therapy on COVID-19 Patients With Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other); Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Andri Maruli Tua Lubis, Head of Research Division RSCM, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: convalescent plasma RSCM-FKUI
Record Dates: First submitted 2020-05-04; First posted 2020-05-08 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: COVID; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- convalescent plasma and standard of care (Experimental)
  Interventions: Biological: Convalescent plasma; Drug: Standard of care
- standard of care (Active Comparator)
  Interventions: Drug: Standard of care

INTERVENTIONS:
Biological: Convalescent plasma — Convalescent plasma of recovered COVID-19 patients (donor)
  Arms: convalescent plasma and standard of care
Drug: Standard of care — According to national or hospital guidelines "COVID-19 Management Protocol"

SUMMARY:
Corona virus disease 2019 (COVID-19) has been declared as a Pandemic by the World Health Organization (WHO). According to WHO report on March 31st 2020, globally COVID-19 have infected over 750,000 people and caused over 36,000 deaths with case fatality rate of 4.85%. In Indonesia, COVID-19 have infected 1,414 people and caused 122 deaths with case fatality rate of 8.63%. In severe cases, COVID-19 causes complications, such as acute respiratory distress syndrome (ARDS), sepsis, septic shock, and multi-organ dysfunction syndrome (MODS), where age and comorbid illnesses as a major factor to these complications. Up to this point there are several promising therapies for COVID-19 but is not yet recommended and in need of further research. The use of convalescent plasma has been approved by the US Food and Drug Administration (FDA) through the scheme of emergency investigational new drug (eIND). This method has been used as the treatment in several outbreak or plague cases over the years, such as the flu epidemic in 1918, polio, measles, mumps, SARS (severe acute respiratory syndrome), EVD (Ebola virus disease) and MERS (middle-eastern respiratory syndrome) and this treatment shows better outcome. Several case report on the use of convalescent plasma for COVID-19 patients with ARDS and mechanical ventilation has been reported and shows promising outcome. Nevertheless, larger and multicenter research need to be done to assess and evaluate the effectiveness and safety of convalescent plasma therapy on for COVID-19 patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than equal to 18 years.
* COVID-19 confirmed by reverse transcriptase-polymerase chain reaction (RT-PCR)
* Having severe pneumonia.
* PAO2 / FIO2 <300.

Exclusion Criteria:

* Contraindication to blood transfusions (fluid overload, history of anaphylaxis of blood products)
* Multiple and severe organ failure, hemodynamically unstable
* Other uncontrolled infections
* Disseminated intravascular coagulation (DIC) which requires a replacement factor/FFP
* Hemodialysis patients or CRRT (continuous renal replacement therapy)
* Active intracranial bleeding
* Significant myocardial ischemia
* Receiving tocilizumab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | up to 28 days
  Proportion of all-cause mortality

SECONDARY OUTCOMES:
Length of stay in intensive care unit | up to 28 days
  Mean length of stay in intensive care unit
Duration of mechanical ventilation | up to 28 days
  Mean duration of mechanical ventilation
Body temperature (degree in Celsius) | Day 1, 3, 5, and 7 after administration of therapy
  Mean change from baseline using time series analysis
The Sequential Organ Failure Assessment (SOFA) Score | Day 1, 3, 5, and 7 after administration of therapy
  Mean change from baseline using time series analysis
PAO2/FIO2 ratio | Day 1, 3, 5, and 7 after administration of therapy
  Mean change from baseline using time series analysis
C-Reactive Protein (CRP) in mg/L | Day 1, 3, 5, and 7 after administration of therapy
  Mean change from baseline using time series analysis
D-Dimer in ng/mL | Day 1, 3, 5, and 7 after administration of therapy
  Mean change from baseline using time series analysis
Procalcitonin in ng/mL | Day 1, 3, 5, and 7 after administration of therapy
  Mean change from baseline using time series analysis
Interleukin 6 (IL-6) in pg/mL | Day 1, 3, 5, and 7 after administration of therapy
  Mean change from baseline using time series analysis
Allergic/ anaphylaxis transfusion reaction | 24 hours post-transfusion
  Number of participants with allergic/ anaphylaxis transfusion reaction
Hemolytic transfusion reaction | 24 hours post-transfusion
  Number of participants with Hemolytic transfusion reaction
Transfusion Related Acute Lung Injury | 24 hours post-transfusion
  Number of participants with Transfusion Related Acute Lung Injury
Transfusion associated Circulatory Overload | 24 hours post-transfusion
  Number of participants with Transfusion associated Circulatory Overload

CONTACTS AND LOCATIONS:
Overall Officials: Andri MT Lubis, MD, PhD, Study Chair — Faculty of Medicine Universitas Indonesia - Dr Cipto Mangunkusumo Hospital
Locations (3):
- Indonesia (3):
  - Dr. Cipto Mangunkusumo General Hospital, Jakarta, DKI Jakarta
  - St. Carolus Hospital, Jakarta, DKI Jakarta
  - Ciputra Hospital CitraRaya, Jakarta, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812
- [Background] Tanne JH. Covid-19: FDA approves use of convalescent plasma to treat critically ill patients. BMJ. 2020 Mar 26;368:m1256. doi: 10.1136/bmj.m1256. No abstract available. PMID 32217555
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] van Griensven J, Edwards T, de Lamballerie X, Semple MG, Gallian P, Baize S, Horby PW, Raoul H, Magassouba N, Antierens A, Lomas C, Faye O, Sall AA, Fransen K, Buyze J, Ravinetto R, Tiberghien P, Claeys Y, De Crop M, Lynen L, Bah EI, Smith PG, Delamou A, De Weggheleire A, Haba N; Ebola-Tx Consortium. Evaluation of Convalescent Plasma for Ebola Virus Disease in Guinea. N Engl J Med. 2016 Jan 7;374(1):33-42. doi: 10.1056/NEJMoa1511812. PMID 26735992
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Zhang W, Du RH, Li B, Zheng XS, Yang XL, Hu B, Wang YY, Xiao GF, Yan B, Shi ZL, Zhou P. Molecular and serological investigation of 2019-nCoV infected patients: implication of multiple shedding routes. Emerg Microbes Infect. 2020 Feb 17;9(1):386-389. doi: 10.1080/22221751.2020.1729071. eCollection 2020. PMID 32065057
- [Background] Rawal G, Yadav S, Kumar R. Acute Respiratory Distress Syndrome: An Update and Review. J Transl Int Med. 2018 Jun 26;6(2):74-77. doi: 10.1515/jtim-2016-0012. eCollection 2018 Jun. PMID 29984201
- [Background] Griffiths MJD, McAuley DF, Perkins GD, Barrett N, Blackwood B, Boyle A, Chee N, Connolly B, Dark P, Finney S, Salam A, Silversides J, Tarmey N, Wise MP, Baudouin SV. Guidelines on the management of acute respiratory distress syndrome. BMJ Open Respir Res. 2019 May 24;6(1):e000420. doi: 10.1136/bmjresp-2019-000420. eCollection 2019. PMID 31258917
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Riviello ED, Kiviri W, Twagirumugabe T, Mueller A, Banner-Goodspeed VM, Officer L, Novack V, Mutumwinka M, Talmor DS, Fowler RA. Hospital Incidence and Outcomes of the Acute Respiratory Distress Syndrome Using the Kigali Modification of the Berlin Definition. Am J Respir Crit Care Med. 2016 Jan 1;193(1):52-9. doi: 10.1164/rccm.201503-0584OC. PMID 26352116
- [Background] Young BE, Ong SWX, Kalimuddin S, Low JG, Tan SY, Loh J, Ng OT, Marimuthu K, Ang LW, Mak TM, Lau SK, Anderson DE, Chan KS, Tan TY, Ng TY, Cui L, Said Z, Kurupatham L, Chen MI, Chan M, Vasoo S, Wang LF, Tan BH, Lin RTP, Lee VJM, Leo YS, Lye DC; Singapore 2019 Novel Coronavirus Outbreak Research Team. Epidemiologic Features and Clinical Course of Patients Infected With SARS-CoV-2 in Singapore. JAMA. 2020 Apr 21;323(15):1488-1494. doi: 10.1001/jama.2020.3204. PMID 32125362
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Qin C, Zhou L, Hu Z, Zhang S, Yang S, Tao Y, Xie C, Ma K, Shang K, Wang W, Tian DS. Dysregulation of Immune Response in Patients With Coronavirus 2019 (COVID-19) in Wuhan, China. Clin Infect Dis. 2020 Jul 28;71(15):762-768. doi: 10.1093/cid/ciaa248. PMID 32161940
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Roback JD, Guarner J. Convalescent Plasma to Treat COVID-19: Possibilities and Challenges. JAMA. 2020 Apr 28;323(16):1561-1562. doi: 10.1001/jama.2020.4940. No abstract available. PMID 32219429
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- See also: Coronavirus disease 2019 Situation Report — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200331-sitrep-71-covid-19.pdf?sfvrsn=4360e92b_4
- See also: Coronavirus disease (COVID-19) in a paucisymptomatic patient: epidemiological and clinical challenge in settings with limited community transmission, Italy, February 2020. — https://www.eurosurveillance.org/content/10.2807/1560-7917.ES.2020.25.11.2000230
- See also: Serological and molecular findings during SARS-CoV-2 infection: the first case study in Finland, January to February 2020 — https://www.eurosurveillance.org/content/10.2807/1560-7917.ES.2020.25.11.2000266